CLINICAL TRIAL: NCT00276107
Title: An Open-Label Trial of the Immunogenicity and Safety of Prevenar (Pneumococcal 7-Valent Conjugate Vaccine [Diphteria CRM197 Protein Conjugate]) in Healthy Infants at 2, 4 and 6 Months of Age
Brief Title: Study Evaluating Prevenar Vaccine in Healthy Infants
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 0887X-101446
Record Dates: First submitted 2006-01-11; First posted 2006-01-12 (Estimated); Last update posted 2009-07-29 (Estimated); Status verified 2009-07

CONDITIONS: Pneumococcal Infections
Keywords: Vaccine; Healthy Infants
MeSH Terms: conditions — Pneumococcal Infections | interventions — Heptavalent Pneumococcal Conjugate Vaccine

INTERVENTIONS:
Biological: Prevenar

SUMMARY:
To determine the immunogenicity of Prevenar in infants immunized at 2, 4 and 6 months of age. To determine the antibody responses to the seven pneumococcal vaccine serotypes one month after second dose and determine the safety of Prevenar in infants immunized at 2,4 and 6 months of age.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female children 2 months of age (42 to 100 days) in good health.
* An informed consent must be signed by a parent or legal guardian following a detailed explanation of participation in the study.
* Infants whose parent(s)/guardian(s) will be available for the entire study period.

Exclusion Criteria:

* Hypersensitivity to any component of the vaccine, including diphtheria toxoid
* Infants with thrombocytopenia or any coagulation disorder that would contraindicate intramuscular injection
* Infants with known or suspected impairment of immunologic functions including HIV or those receiving immunosuppressive therapy.

Other exclusions apply.

Ages: 42 Days to 100 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200
Dates: Start 2004-12; Study Completion 2005-12

PRIMARY OUTCOMES:
To determine the immunogenicity of Prevenar in infants immunized at 2, 4 and 6 months of age

SECONDARY OUTCOMES:
To determine the antibody responses to the seven pneumococcal vaccine serotypes after second dose and to determine the safety of Prevenar in infants immunized at 2, 4 and 6 months of age

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer